CLINICAL TRIAL: NCT07063563
Title: Effect of Rehabilitation at Moderate Altitude on Airway Resistance Measured With Forced Oscillation Technique in Patients With COPD
Brief Title: Effect of Rehabilitation at Moderate Altitude on Airway Resistance Measured With Forced Oscillation Technique in COPD-patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Switzerland University of Applied Sciences (Other)
Collaborators: National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov (Other Government); University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: inRehaExO2_FOT
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: COPD
Keywords: Oxygen; Exercise; Rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normoxia (Sham Comparator): Sham air (ambient air) (5l/min) will be applied with the oxygen concentrator EverFlo TM via nasal cannula
  Interventions: Other: ambiant air
- Hyperoxia (Active Comparator): Standardized supplemental oxygen therapy (SSOT) at 5 L/min will be delivered using the EverFlo™ oxygen concentrator via nasal cannula during training.
  Interventions: Other: Oxygen
- Hypoxia (Experimental): This group will train at moderate altitude
  Interventions: Other: ambiant air

INTERVENTIONS:
Other: ambiant air — Standard ambiant air will be breathed during endurance training. ambiant air
  Arms: Hypoxia
Other: Oxygen — SSOT and sham air (5l/min) will be applied with the oxygen concentrator EverFloTM via nasal cannula during training
  Arms: Hyperoxia
Other: ambiant air — Standard ambiant air will be breathed during endurance training. ambiant air
  Arms: Normoxia

SUMMARY:
Airway resistance will be measured using the forced oscillation technique (FOT). The parameters Rrs, Xrs, and ∆Xrs will be compared before and after a pulmonary rehabilitation cycle at moderate altitude. Additionally, the differences between low and moderate altitude will also be examined.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Stable clinical condition for >3 weeks (e.g., no exacerbations)
* Resting SpO₂ ≥88% and exercise-induced hypoxemia defined as a drop in SpO₂ of ≥4% and/or a level below 90% during the 6MWT
* Informed consent documented by signature

Exclusion Criteria:

* Severe daytime resting hypoxemia (SpO₂ <88%)
* Long-term oxygen therapy
* Unstable clinical condition requiring adjustment of pharmacological or other treatment modalities, need for intensive care, or presence of relevant severe comorbidities
* Inability to comply with study procedures (e.g., due to language barriers, psychological disorders, neurological or orthopedic impairments, walking disability, or inability to ride a bicycle)
* Women who are pregnant or breastfeeding
* Enrolment in another clinical trial involving active treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-07-23 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
1. Change in Rrs (Respiratory System Resistance) before and after rehabilitation cycle | baseline to 3 weeks
  Rrs will be measured using the forced oscillation technique (FOT) in cmH₂O·s/L. Values will be assessed before and after the pulmonary rehabilitation cycle at moderate altitude

SECONDARY OUTCOMES:
Change in Xrs (Respiratory System Reactance) compared before and after the pulmonary rehabilitation. | baseline to 3 weeks
  Xrs will be measured using FOT in cmH₂O·s/L. Values will be compared before and after the pulmonary rehabilitation
Change in ∆Xrs (Difference in Reactance) before and after rehabilitation | baseline to 3 weeks
  ∆Xrs will be calculated as the difference between inspiratory and expiratory Xrs values, measured in cmH₂O·s/L, before and after rehabilitation.
Change in Rrs, Xrs and ∆Xrs from low to moderate altitude | From baseline at low altitude to transfer to moderate altitude at 3 days

CONTACTS AND LOCATIONS:
Locations (2):
- National center for cardiology and internal medicine, Bishkek, Kyrgyzstan, Kyrgyzstan
- Eastern Switzerland University of Applied Sciences, Sankt Gallen, Canton of St. Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No
individual patient data will be shared upon personal request to the corresponding author